CLINICAL TRIAL: NCT01208129
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter, Parallel Group Study of the Safety and Efficacy of NAB001 in the Treatment of Mild to Moderate Distal Subungual Onychomycosis of the Toenails for 52 Weeks
Brief Title: Safety and Efficacy of NAB001 in the Treatment of Mild to Moderate Onychomycosis of the Toenails
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0903
Record Dates: First submitted 2010-09-20; First posted 2010-09-23 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Onychomycosis
Keywords: toenail fungus; onychomycosis; nail infection
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug (Experimental)
  Interventions: Drug: NAB001
- Vehicle alone (Placebo Comparator)
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: NAB001 — nail lacquer, once daily, 52 weeks
  Arms: Active drug
Drug: Placebo control — nail lacquer, once daily, 52 weeks
  Arms: Vehicle alone

SUMMARY:
The objectives of this study are to assess the safety of NAB001 for topical treatment of mild to moderate distal onychomycosis of the toenails over 52 weeks and to compare the efficacy of NAB001 to vehicle alone at the end of the study (Week 56) after treating for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate fungal infection of the toenail as assessed by study doctor
* koh positive & dermatophyte culture positive at Visit 1
* general good health as assessed by study doctor

Exclusion Criteria:

* severe fungal toenail infection
* prior use of antifungal drugs (wash-out allowed, duration varies on class)
* significant confounding conditions as assessed by study doctor
* pregnancy/lactation
* must forego nail salon procedures during study for at least ~60 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Complete cure rate at Week 56. Complete cure defined as clinically clear nail and mycological cure. | Week 56 after 52 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects with effective treatment at week 56. Effective treatment defined as mycological cure and an IGA of 0 or 1 (clear or almost clear). | Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Kent Allenby, MD, Study Director — Promius Pharma; Joanne Fraser, PhD, Study Director — Promius Pharma
Locations (25):
- United States (25):
  - Radiant Research, Inc., Tucson, Arizona
  - Associated Foot & Ankle Specialists, LLC, Phoenix, Arkansas
  - Family Foot Health Center, Rogers, Arkansas
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - UCSF Dermatology Research, San Francisco, California
  - Avail Clinical Research, DeLand, Florida
  - North Florida Dermatology Association, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - Lake Washington Foot and Ankle Center, Melbourne, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Department of Veteran's Affairs, Minneapolis, Minnesota
  - Pinkas Lebovits, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - Care Plus Podiatry, PC, Wading River, New York
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Radiant Research, Inc., Greer, South Carolina
  - The Skin Wellness Center, PC, Knoxville, Tennessee
  - Research Across America, Plano, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Coastal Podiatry, Inc., Virginia Beach, Virginia
  - Madison Skin and Research, Inc., Madison, Wisconsin